CLINICAL TRIAL: NCT01494857
Title: Open-Label, Non-Randomized, Single Patient Group, Multi-Center Study to Evaluate the Efficacy and Safety of Adalimumab for the Induction of Clinical Response in Moderately to Severely Active Ulcerative Colitis
Brief Title: Efficacy and Safety of Adalimumab for the Induction of Clinical Response in Ulcerative Colitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Timna Naftali, Principal Investigator, Clalit Health Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KHK - AD001; A13-675 (Other Grant/Funding Number: Abbott)
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; biological treatment; anti-TNF
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab (Experimental): Adalimumab 40 mg
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Adalimumab 40 mg from 4 to 1 injection once in two weeks. Total Treatment period - 10 weeks.
  Other Names: Brand name - Humira (Abbott Pharmaceuticals)

SUMMARY:
The purpose of this study is to assess the clinical benefit and tolerability of adalimumab, a fully human monoclonal antibody to tumor necrosis factor α (TNF- α), in patients with ulcerative colitis (UC) naive to treatment with biologics.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is one of the two primary forms of idiopathic inflammatory bowel disease (IBD). Recent studies have shown that TNF- α may play a major role in the etiopathogenesis of UC, justifying the use of anti-TNF-α therapies. Adalimumab is an immunoglobulin G1 that specifically binds to TNF-α, and neutralizes its function; it also modulates the biological response, induced and regulated by TNF-α.

Conventional UC therapy quite commonly does not bring satisfactory results; therefore, interest in new treatment methods has been growing recently. Biological therapy is a highly promising prospect, since it enables to discontinue the use of glucocorticosteroids and immunosuppressives or their dose reduction, shortens the hospitalization period, allows to avoid surgical treatment, extends the clinical response, the remission period and improves the patient's quality of life.

Thus, the present study assesses the clinical response of active ulcerative colitis to adalimumab treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age.
2. Diagnosis of ulcerative colitis for greater than 90 days prior to Baseline.
3. Diagnosis of active UC confirmed by colonoscopy with biopsy or flexible sigmoidoscopy with biopsy during the Screening Period, with exclusion of infection.
4. Active UC with a Mayo score of 6 to 12 points and endoscopy subscore of 2 to 3 points, despite concurrent treatment with at least 1 of the following (oral corticosteroids or immunosuppressants or both as defined below):

   * Stable oral corticosteroid dose (prednisone dose of >= 20 mg/day or equivalent) for at least 14 days prior to Baseline or stable oral corticosteroid dose (prednisone of < 20 mg/day) for at least 40 days prior to Baseline, and/or
   * At least a consecutive 90 day course of azathioprine or 6-mercaptopurine (6 MP) prior to Baseline, with a dose of azathioprine >= 1.5 mg/kg/day or 6 MP >= 1 mg/kg/day (rounded to the nearest available tablet formulation), or a dose that is the highest tolerated by the participant (e.g., due to leukopenia, elevated liver enzymes, nausea) during that time. Participant was to be on a stable dose for at least 28 days prior to Baseline.
5. Concurrent therapy was not required for participants who were previously treated with corticosteroids or immunosuppressants (azathioprine or 6-MP) during the previous 5 years and, in the judgment of the investigator, have failed to respond to or could not tolerate their treatment.
6. Has to be able to self-administer subcutaneous injections or has caregiver who can reliably administer subcutaneous injections.
7. Has to be able and willing to give written informed consent and to comply with the requirements of this study protocol.

Exclusion Criteria:

1. History of subtotal colectomy with ileorectostomy or colectomy with ileoanal pouch, Koch pouch, or ileostomy for UC or is planning bowel surgery.
2. Received previous treatment with adalimumab or previous participation in an adalimumab clinical study.
3. Received cyclosporine, tacrolimus, or mycophenolate mofetil, within 30 days prior to Baseline.
4. Received intravenous corticosteroids within 14 days prior to Screening or during the Screening Period.
5. Received therapeutic enema or suppository, other than required for endoscopy, within 14 days prior to the Screening endoscopy and during the remainder of Screening Period.
6. Current diagnosis of fulminant colitis and/or toxic megacolon.
7. Subject with disease limited to the rectum (ulcerative proctitis).
8. Current diagnosis of indeterminate colitis.
9. Current diagnosis and/or history of Crohn's disease.
10. Currently receiving total parenteral nutrition (TPN).
11. Subject using aminosalicylates for less than 90 days prior to Baseline or not on a stable dose for at least 28 days prior to Baseline or discontinued use within 28 days of Baseline.
12. Subject with positive Clostridium difficile (C. difficile) stool assay.
13. Subject who has previously used infliximab or any anti-TNF agent within 56 days of Baseline.
14. Subject who has previously used infliximab or any anti-TNF agent and has not clinically responded at any time ("primary non-responder") unless subject experienced a treatment limiting reaction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with clinical response per Mayo Score, at Week 12 | week 12

SECONDARY OUTCOMES:
Proportion of subjects with remission per Mayo Score at Week 12. | week 12

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Sherutey Briuth Clalit / Clalit HMO, Herzlyia
  - Lev Talpiot Clinic, Clalit health Services, Jerusalem
  - Zevulun Clinic, Clalit Health Services, Kiryat Bialik